CLINICAL TRIAL: NCT03941093
Title: A Phase 3, Randomized, Double-Blind Study of Pamrevlumab or Placebo in Combination With Either Gemcitabine Plus Nab-paclitaxel or FOLFIRINOX as Neoadjuvant Treatment in Patients With Locally Advanced, Unresectable Pancreatic Cancer
Brief Title: Evaluation of Efficacy and Safety of Neoadjuvant Treatment With Pamrevlumab in Combination With Chemotherapy (Either Gemcitabine Plus Nab-paclitaxel or FOLFIRINOX) in Participants With Locally Advanced, Unresectable Pancreatic Cancer
Acronym: LAPIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyntra Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FGCL-3019-087
Record Dates: First submitted 2019-05-02; First posted 2019-05-07 (Actual); Results first posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-09

CONDITIONS: Pancreatic Cancer Non-resectable
Keywords: locally advanced pancreatic cancer; unresectable pancreatic cancer
MeSH Terms: interventions — pamrevlumab; Gemcitabine; 130-nm albumin-bound paclitaxel; folfirinox; Albumin-Bound Paclitaxel; Leucovorin; Irinotecan; Fluorouracil

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1 ratio to one of the two study treatment arms; pamrevlumab with G/NP or FOLFIRINOX or placebo with G/NP or FOLFIRINOX.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Pamrevlumab + Gemcitabine + Nab-paclitaxel or Pamrevlumab + FOLFIRINOX
  Interventions: Drug: Pamrevlumab + Gemcitabine + Nab-paclitaxel or Pamrevlumab + FOLFIRINOX
- Arm B (Placebo Comparator): Placebo + Gemcitabine + Nab-paclitaxel or Placebo + FOLFIRINOX
  Interventions: Drug: Placebo + Gemcitabine + Nab-paclitaxel or Placebo + FOLFIRINOX

INTERVENTIONS:
Drug: Pamrevlumab + Gemcitabine + Nab-paclitaxel or Pamrevlumab + FOLFIRINOX — Drug: Pamrevlumab is administered on Days 1, 8 and 15 of Treatment Cycle 1 and on Day 1 and 15 of each subsequent treatment cycle via IV infusion.
  Drug: Gemcitabine is administered on Days 1, 8 and 15 of each 28 day treatment cycle via IV infusion.
  Drug: Nab-paclitaxel is administered on Days 1, 8 and 15 of each 28 day treatment cycle via IV infusion.
  Drug: FOLFIRINOX is a combination of several agents administered on Days 1 and 15 of each 28 day treatment cycle via IV infusion. The specific agents are Oxaliplatin, Folinic Acid, Irinotecan, and Fluorouracil.
  Other Names: FG-3019; Gemzar; Abraxane; Eloxitan; Leucovorin; Camptosar; 5-Fluracil; Efudex
  Arms: Arm A
Drug: Placebo + Gemcitabine + Nab-paclitaxel or Placebo + FOLFIRINOX — Drug: Placebo is administered on Days 1, 8 and 15 of Treatment Cycle 1 and on Day 1 and 15 of each subsequent treatment cycle via IV infusion.
  Drug: Gemcitabine is administered on Days 1, 8 and 15 of each 28 day treatment cycle via IV infusion.
  Drug: Nab-paclitaxel is administered on Days 1, 8 and 15 of each 28 day treatment cycle via IV infusion.
  Drug: FOLFIRINOX is a combination of several agents administered on Days 1 and 15 of each 28 day treatment cycle via IV infusion. The specific agents are Oxaliplatin, Folinic Acid, Irinotecan, and Fluorouracil.
  Other Names: Gemzar; Abraxane; Eloxitan; Leucovorin; Camptosar; 5-Fluracil; Efudex
  Arms: Arm B

SUMMARY:
This is a Phase 3, randomized, double-blind trial to evaluate the efficacy and safety of neoadjuvant treatment with pamrevlumab or placebo in combination with either gemcitabine plus nab-paclitaxel (G/NP) or FOLFIRINOX in the treatment of participants with locally advanced, unresectable pancreatic cancer.

DETAILED DESCRIPTION:
Participants will be randomized in a 1:1 ratio to one of the two study treatment arms; pamrevlumab with either G/NP or FOLFIRINOX, placebo with G/NP or FOLFIRINOX.

Each participant may receive up to 6 cycles of treatment (each treatment cycle is 28 days). Tumor tissue will be collected during resection to determine surgical outcome and for biomarker analysis. Tumor response will be evaluated by changes in CT scan, FDG-PET, CA 19-9, and NCCN® guidelines.

All participants randomized will have a safety follow-up visit approximately 28 days after the last dose of study treatment and a final safety follow-up phone call at approximately 60 days after the last dose.

Participants who complete study treatment will be evaluated for surgical exploration for possible R0 or R1 resection. Surgery will occur at least 4 weeks after the last dose (allowing for a wash-out period from treatment) and only after receipt of the recommendation from the central review board with regards to surgical eligibility. Surgery will occur no longer than 8 weeks after the last dose. Participants who undergo surgery will be evaluated for surgical complications for at least an additional 90 days following discharge from surgery.

Participants who are ineligible for surgical exploration (i.e. participants who did not complete study treatment or do not meet any of the protocol defined criteria or had a contraindication to surgery) will continue in the Follow-up period and receive treatment as per standard of care (SOC) for each institution.

All participants will be followed for disease progression (if not previously detected) or recurrence following resection (local progression or metastatic disease). Participants will also be followed for any additional anti-cancer therapy received for their pancreatic cancer. All participants will be followed for survival (until death) or until the last participant to complete treatment reaches 18 months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and sign informed consent; be willing to comply with study procedures, including surgery
2. Age ≥ 18 years
3. Be a male, or non-pregnant and non-lactating female
4. Negative serum B-hCG pregnancy test at screening for women of childbearing potential
5. Male participants with partners of childbearing potential and female participants of childbearing potential are required to use highly effective contraception methods during the conduct of the study and for 6 months after the last dose of study drug
6. Histologically or cytologically proven diagnosis of pancreatic ductal adenocarcinoma (PDAC)
7. Locally advanced pancreatic cancer considered unresectable according to NCCN Guidelines® Version 2.2018 as determined by central imaging
8. Measurable disease as defined by RECIST 1.1 criteria as determined by central imaging
9. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
10. Adequate liver function: aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <2.5 x upper limit of normal (ULN), alkaline phosphatase <2.5 x ULN, and bilirubin ≤1.5 x ULN or in participants with biliary stenting ≤2.0 x ULN
11. Adequate bone marrow function: platelets >100,000 cells/mm3, hemoglobin >9.0 g/dl and absolute neutrophil count (ANC) >1,500 cells/mm3
12. Adequate renal function: creatinine < 1.5 x ULN, creatinine clearance ≥ 30 mL/min
13. Less than grade 2 pre-existing peripheral neuropathy (per CTCAE)

Exclusion Criteria:

1. Prior chemotherapy or radiation for pancreatic cancer
2. Previous (within the past 3 years) or concurrent malignancy diagnosis except non-melanoma skin cancer and in situ carcinomas (excluding in situ breast cancer)
3. Major surgery within 4 weeks prior to signing informed consent form. Biliary stents are permitted.
4. History of allergy or hypersensitivity to human, humanized or chimeric monoclonal antibodies
5. History of allergy or hypersensitivity to any of the chemotherapy agents being prescribed or their excipients
6. Any medical or surgical condition that may place the participant at increased risk while on study
7. Any condition potentially decreasing compliance to study procedures
8. Exposure to another investigational drug within 28 days of first dosing visit, or 5 half-lives of the investigational drug (whichever is longer)
9. Uncontrolled intercurrent illness including, but not limited to, ongoing or active systemic infections, symptomatic congestive heart failure, unstable angina pectoris, clinically significant cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
10. Documented history of drug or alcohol abuse within 6 months of signing informed consent
11. Any medical condition that, in the opinion of the investigator, may pose a safety risk to a participant in this trial, may confound the assessment of safety and efficacy, or may interfere with study participation
12. Participants with a history of interstitial pulmonary disease, hepatitis C virus (HCV), hepatitis B virus (HBV) or human immunodeficiency virus (HIV) infection
13. Participants who have been administered a live vaccine within 4 weeks prior to the first administration of therapy
14. Participants who cannot stop chronic medications that inhibit or induce cytochrome P (CYP) 2C8 or CYP3A4
15. Participants with poorly controlled comorbid conditions, including; congestive heart failure (CHF), chronic obstructive pulmonary disease (COPD), uncontrolled diabetes mellitus (DM) or neurologic disorders (not acutely related to pancreatic cancer) or limited function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2024-06-11 (Actual); Study Completion 2024-06-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (90):
- United States (32):
  - St. Joseph's Hospital and Medical Cancer Center, Phoenix, Arizona
  - UC San Diego Moores Cancer Center, La Jolla, California
  - UCLA, Los Angeles, California
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - Elmhurst Memorial Hospital - Nancy W. Knowles Cancer Center, Elmhurst, Illinois
  - Edward Cancer Center, Naperville, Illinois
  - Indiana University Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - University of Kansas Hospital, Westwood, Kansas
  - Norton Cancer Institute, Audubon Hospital Campus, Louisville, Kentucky
  - Maine Health Cancer Care, South Portland, Maine
  - University of Massachusetts, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Saint Luke's Hospital, Kansas City, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - New Mexico Cancer Care Alliance, Albuquerque, New Mexico
  - NYU Langone Health, New York, New York
  - Stony Brook University, Stony Brook, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Reading Hospital McGlinn Cancer Institute, West Reading, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Baylor Scott & White Medical Center, Temple, Texas
  - Renovatio Clinic, The Woodlands, Texas
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - West Virginia University, Morgantown, West Virginia
- Austria (2):
  - Medizinische Universität Wien, Vienna
  - Klinikum Wels-Grieskirchen GmbH, Wels
- CUB Hôpital Erasme, Brussels, Belgium
- Canada (4):
  - The Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Princess Margaret Cancer Centre/University Health Network, Toronto, Ontario
  - McGill University Health Center, Montreal, Quebec
- China (8):
  - Peking Union Medical College Hospital, Dongcheng, Beijing Municipality
  - Union Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - The First Affiliated Hospital Of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Huashan Hospital affiliated with Fudan University, Jing’an, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu
  - Jiangsu Province Hospital, Nanjing
  - Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai
  - Xinhua Hospital Affiliated to Shanghai Jiaotong University School Of Medicine, Shanghai
- France (10):
  - CHRU Jean Minjoz, Besançon
  - CHU Estaing, Clermont-Ferrand
  - Hopital BEAUJON, Clichy
  - Centre Georges-François Leclerc, Dijon
  - CHU Grenoble Alpes, La Tronche
  - Centre Léon Bérard, Lyon
  - Hôpital Edouard Herriot, Lyon
  - Groupe Hospitalier Pitié Salpêtrière, Paris
  - Haut-Lévêque, Pessac
  - Institut de Cancérologie de l'Ouest Pays de Loire, Saint-Herblain
- Germany (4):
  - Medizinische Klinik mit Schwerpunkt Hämatologie, Onkologie und Tumorimmunologie, Berlin
  - Technische Universität Dresden, Medizinische Klinik und Poliklinik I, Dresden
  - Klinikum der Universität München, Medizinische Klinik und Poliklinik III, München
  - Klinikum rechts der Isar der Technischen Universität München, München
- Israel (4):
  - Shamir Medical center Asaf Harofeh, Be’er Ya‘aqov
  - Hadassah University Hospital Ein Kerem, Jerusalem
  - Meir Medical center, Kfar Saba
  - Rabin Medical Center, Petah Tikva
- Italy (7):
  - Instituto Scientifico Romagnolog per lo Studio e la Cura dei Tumori, Meldola
  - IRCCS Ospedale San Raffaele, Milan
  - Istituto Europeo di Oncologia, Milan
  - Grande Ospedale Metropolitano Niguarda, Oncologia Medica Falck, Milan
  - AOU Federico II, Napoli
  - Istituto Clinico Humanitas, Rozzano
  - CRC di Verona, Verona
- South Korea (7):
  - Seoul National University Budang Hospital, Seongnam-si, Geyonggi-do
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Chonnam National University Hwasun Hospital, Hwasun, Jeollanam-do
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Spain (9):
  - Alvaro Cunqueiro Hospital, Vigo, Pontevedra
  - Hospital Universitaro Vall D'Hebron, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Institut Catalá d'Oncologia (ICO Girona). Hospital Dr. Josep Trueta, Girona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - MD Anderson Cancer Center, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- United Kingdom (2):
  - University College London Hospitals NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Link to sponsor website — http://www.fibrogen.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized in a 1:1 ratio to one of the 2 study treatment arms: Pamrevlumab with Gemcitabine/Nab-paclitaxel or FOLFIRINOX or Placebo with Gemcitabine/Nab-paclitaxel or FOLFIRINOX.
Groups:
- Pamrevlumab + Gemcitabine/Nab-paclitaxel or FOLFIRINOX: Participants received pamrevlumab in combination with one chemotherapy treatment regimen (gemcitabine plus nab-paclitaxel or FOLFIRINOX) over a 28-day cycle, for up to 6 cycles. Pamrevlumab was administered on Days 1, 8 and 15 of Treatment Cycle 1 and on Day 1 and 15 of each subsequent treatment cycle via intravenous (IV) infusion. Nab-paclitaxel was administered on Days 1, 8 and 15 of each 28-day treatment cycle via IV infusion. Gemcitabine was administered on Days 1, 8 and 15 of each 28-day treatment cycle via IV infusion. FOLFIRINOX was a combination of several agents administered on Days 1 and 15 of each 28-day treatment cycle via IV infusion. The specific agents were oxaliplatin, folinic acid, irinotecan, and fluorouracil.
- Placebo + Gemcitabine/Nab-paclitaxel or FOLFIRINOX: Participants received pamrevlumab matched placebo in combination with one chemotherapy treatment regimen (gemcitabine plus nab-paclitaxel or FOLFIRINOX) over a 28-day cycle, for up to 6 cycles. Placebo was administered on Days 1, 8 and 15 of Treatment Cycle 1 and on Day 1 and 15 of each subsequent treatment cycle via IV infusion. Nab-paclitaxel was administered on Days 1, 8 and 15 of each 28-day treatment cycle via IV infusion. Gemcitabine was administered on Days 1, 8 and 15 of each 28-day treatment cycle via IV infusion. FOLFIRINOX was a combination of several agents administered on Days 1 and 15 of each 28-day treatment cycle via IV infusion. The specific agents were oxaliplatin, folinic acid, irinotecan, and fluorouracil.
Period: Overall Study
Arm/Group | Pamrevlumab + Gemcitabine/Nab-paclitaxel or FOLFIRINOX | Placebo + Gemcitabine/Nab-paclitaxel or FOLFIRINOX
Started | 143 | 141
Received At Least 1 Dose of Study Drug | 142 | 141
Completed | 134 | 134
Not Completed | 9 | 7
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 9 | 6

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population included all randomized participants regardless of whether or not study treatment was received.
Groups:
- Pamrevlumab + Gemcitabine/Nab-paclitaxel or FOLFIRINOX: Participants received pamrevlumab in combination with one chemotherapy treatment regimen (gemcitabine plus nab-paclitaxel or FOLFIRINOX) over a 28-day cycle, for up to 6 cycles. Pamrevlumab was administered on Days 1, 8 and 15 of Treatment Cycle 1 and on Day 1 and 15 of each subsequent treatment cycle via IV infusion. Nab-paclitaxel was administered on Days 1, 8 and 15 of each 28-day treatment cycle via IV infusion. Gemcitabine was administered on Days 1, 8 and 15 of each 28-day treatment cycle via IV infusion. FOLFIRINOX was a combination of several agents administered on Days 1 and 15 of each 28-day treatment cycle via IV infusion. The specific agents were oxaliplatin, folinic acid, irinotecan, and fluorouracil.
- Total: Total of all reporting groups
Arm/Group | Pamrevlumab + Gemcitabine/Nab-paclitaxel or FOLFIRINOX | Placebo + Gemcitabine/Nab-paclitaxel or FOLFIRINOX | Total
Number analyzed (Participants) | 143 | 141 | 284
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (9.54) | 64.5 (9.60) | 64.5 (9.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 72 | 133
  Male | 82 | 69 | 151
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 2 | 12
  Not Hispanic or Latino | 122 | 124 | 246
  Unknown or Not Reported | 11 | 15 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 25 | 35 | 60
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 96 | 79 | 175
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 17 | 20 | 37

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival was defined as the time from date of randomization to date of death due to any cause. Overall survival was calculated using the Kaplan-Meier method.
Time Frame: Up to approximately 5 years
Population: The ITT population included all randomized participants regardless of whether or not study treatment was received.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pamrevlumab + Gemcitabine/Nab-paclitaxel or FOLFIRINOX | Placebo + Gemcitabine/Nab-paclitaxel or FOLFIRINOX
Number analyzed (Participants) | 143 | 141
months | 17.25 [15.47 to 18.89] | 17.94 [14.59 to 20.34]
Statistical Analysis 1: Comparison: Pamrevlumab + Gemcitabine/Nab-paclitaxel or FOLFIRINOX vs Placebo + Gemcitabine/Nab-paclitaxel or FOLFIRINOX; Test type: Other; p = 0.5487, Stratified Log Rank Test; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.83 to 1.41]

2. Secondary Outcome: Event-free Survival (EFS)
Description: The EFS endpoint was a composite time-to-event endpoint. The event being analyzed ('treatment failure') was defined as the earliest occurrence of: a) failure to achieve disease-free status locally after completion of neoadjuvant treatment and/or after surgery (that is, resection failure or progression that precludes surgery); b) local or distant recurrence, or c) death. The EFS was calculated using the Kaplan-Meier method.
Time Frame: Up to approximately 5 years
Population: The ITT population included all randomized participants regardless of whether or not study treatment was received.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pamrevlumab + Gemcitabine/Nab-paclitaxel or FOLFIRINOX | Placebo + Gemcitabine/Nab-paclitaxel or FOLFIRINOX
Number analyzed (Participants) | 143 | 141
months | 5.72 [5.59 to 6.01] | 5.78 [5.62 to 6.37]

3. Secondary Outcome: Progression-free Survival (PFS) as Assessed Using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Description: The PFS was defined as time from date of randomization until disease progression or death due to any cause, whichever occurred first. PFS was calculated using the Kaplan-Meier method. Progression was defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of at least 5 millimeters (mm). Unequivocal progression of existing non-target lesions and the appearance of one or more new lesions was also considered progression.
Time Frame: Up to approximately 5 years
Population: The ITT population included all randomized participants regardless of whether or not study treatment was received.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pamrevlumab + Gemcitabine/Nab-paclitaxel or FOLFIRINOX | Placebo + Gemcitabine/Nab-paclitaxel or FOLFIRINOX
Number analyzed (Participants) | 143 | 141
months | 9.36 [7.75 to 11.79] | 9.40 [7.69 to 10.84]

4. Secondary Outcome: Number of Participants With Best Overall Objective Response as Assessed Using RECIST v1.1
Description: Best overall objective response was defined as a complete response (CR) or partial response (PR). CR was defined as disappearance of all target or non-target lesions and normalization of tumor marker level (for non-target lesions), any pathological lymph nodes (whether target or non-target) must have reduced in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to approximately 5 years
Population: The ITT population included all randomized participants regardless of whether or not study treatment was received.
Measure: Count of Participants; unit: Participants
Arm/Group | Pamrevlumab + Gemcitabine/Nab-paclitaxel or FOLFIRINOX | Placebo + Gemcitabine/Nab-paclitaxel or FOLFIRINOX
Number analyzed (Participants) | 143 | 141
Participants | 43 | 64

ADVERSE EVENTS:
Time Frame: Up to approximately 5 years
Description: Per planned analysis all-cause mortality data were collected and reported for all randomized participants. Adverse events (serious and other) were collected and reported for all randomized participants who received study drug.
Arm/Group | Pamrevlumab + Gemcitabine/Nab-paclitaxel or FOLFIRINOX | Placebo + Gemcitabine/Nab-paclitaxel or FOLFIRINOX
All-Cause Mortality (participants affected / at risk) | 118/143 | 112/141
Serious Adverse Events (participants affected / at risk) | 75/142 | 62/141
Other Adverse Events (participants affected / at risk) | 139/142 | 140/141
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pamrevlumab + Gemcitabine/Nab-paclitaxel or FOLFIRINOX (N=142) | Placebo + Gemcitabine/Nab-paclitaxel or FOLFIRINOX (N=141)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 2
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Hydrocele (Congenital, familial and genetic disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 3
Colitis (Gastrointestinal disorders) | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 3
Vomiting (Gastrointestinal disorders) | 3 | 6
Nausea (Gastrointestinal disorders) | 2 | 4
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Ascites (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Duodenal obstruction (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 2
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Jejunal perforation (Gastrointestinal disorders) | 1 | 0
Obstruction gastric (Gastrointestinal disorders) | 1 | 0
Varices oesophageal (Gastrointestinal disorders) | 1 | 0
Abdominal adhesions (Gastrointestinal disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Pancreatic fistula (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 2
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 5 | 6
Asthenia (General disorders) | 3 | 0
Death (General disorders) | 1 | 0
Hypothermia (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 1
Cholangitis (Hepatobiliary disorders) | 7 | 8
Biliary obstruction (Hepatobiliary disorders) | 3 | 5
Cholecystitis (Hepatobiliary disorders) | 2 | 0
Gallbladder rupture (Hepatobiliary disorders) | 2 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 2 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 1
Malignant biliary obstruction (Hepatobiliary disorders) | 1 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 1
Hepatic cytolysis (Hepatobiliary disorders) | 0 | 1
Liver injury (Hepatobiliary disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1
Sepsis (Infections and infestations) | 7 | 1
Pneumonia (Infections and infestations) | 5 | 4
Liver abscess (Infections and infestations) | 2 | 3
Pneumocystis jirovecii pneumonia (Infections and infestations) | 2 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Biliary tract infection (Infections and infestations) | 1 | 0
Catheter site infection (Infections and infestations) | 1 | 0
Cholangitis infective (Infections and infestations) | 1 | 0
Cholecystitis infective (Infections and infestations) | 1 | 3
Clostridium difficile infection (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 0
Parainfluenzae virus infection (Infections and infestations) | 1 | 0
Post procedural infection (Infections and infestations) | 1 | 1
Septic shock (Infections and infestations) | 1 | 1
Tongue fungal infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
COVID-19 (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Streptococcal bacteraemia (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Anastomotic complication (Injury, poisoning and procedural complications) | 0 | 1
Post procedural fever (Injury, poisoning and procedural complications) | 0 | 1
Post procedural fistula (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 2
Platelet count decreased (Investigations) | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 3 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 2
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Device occlusion (Product Issues) | 1 | 2
Anxiety disorder (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 4 | 2
Renal injury (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Pseudocellulitis (Skin and subcutaneous tissue disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 2
Hypertension (Vascular disorders) | 0 | 2
Shock haemorrhagic (Vascular disorders) | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pamrevlumab + Gemcitabine/Nab-paclitaxel or FOLFIRINOX (N=142) | Placebo + Gemcitabine/Nab-paclitaxel or FOLFIRINOX (N=141)
Fatigue (General disorders) | 84 | 76
Diarrhoea (Gastrointestinal disorders) | 81 | 90
Nausea (Gastrointestinal disorders) | 68 | 73
Anaemia (Blood and lymphatic system disorders) | 54 | 67
Alopecia (Skin and subcutaneous tissue disorders) | 53 | 57
Neutrophil count decreased (Investigations) | 51 | 56
Decreased appetite (Metabolism and nutrition disorders) | 50 | 48
Oedema peripheral (General disorders) | 44 | 52
Constipation (Gastrointestinal disorders) | 38 | 39
Vomiting (Gastrointestinal disorders) | 38 | 40
Platelet count decreased (Investigations) | 36 | 43
Abdominal pain (Gastrointestinal disorders) | 34 | 36
Neutropenia (Blood and lymphatic system disorders) | 31 | 30
Neuropathy peripheral (Nervous system disorders) | 30 | 26
Pyrexia (General disorders) | 30 | 30
Asthenia (General disorders) | 27 | 27
Stomatitis (Gastrointestinal disorders) | 25 | 25
White blood cell count decreased (Investigations) | 24 | 28
Dysgeusia (Nervous system disorders) | 23 | 26
Peripheral sensory neuropathy (Nervous system disorders) | 23 | 29
Alanine aminotransferase increased (Investigations) | 19 | 19
Weight decreased (Investigations) | 19 | 18
Hypokalaemia (Metabolism and nutrition disorders) | 18 | 33
Rash (Skin and subcutaneous tissue disorders) | 18 | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 18 | 23
Aspartate aminotransferase increased (Investigations) | 17 | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17 | 18
Paraesthesia (Nervous system disorders) | 17 | 18
Abdominal pain upper (Gastrointestinal disorders) | 16 | 15
Hypotension (Vascular disorders) | 16 | 13
Insomnia (Psychiatric disorders) | 16 | 20
Headache (Nervous system disorders) | 15 | 18
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 | 18
Hypomagnesaemia (Metabolism and nutrition disorders) | 14 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 14 | 17
Abdominal distension (Gastrointestinal disorders) | 13 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 17
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 12 | 14
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 12 | 12
Dyspepsia (Gastrointestinal disorders) | 11 | 6
Chills (General disorders) | 10 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 21
Dry mouth (Gastrointestinal disorders) | 10 | 6
Fall (Injury, poisoning and procedural complications) | 10 | 7
Blood creatinine increased (Investigations) | 9 | 4
Dehydration (Metabolism and nutrition disorders) | 9 | 8
Dizziness (Nervous system disorders) | 9 | 22
Flatulence (Gastrointestinal disorders) | 9 | 6
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 9 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 9 | 9
Blood alkaline phosphatase increased (Investigations) | 8 | 9
Dry skin (Skin and subcutaneous tissue disorders) | 8 | 6
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 8 | 5
Haemorrhoids (Gastrointestinal disorders) | 7 | 10
Hypoalbuminaemia (Metabolism and nutrition disorders) | 7 | 14
Anxiety (Psychiatric disorders) | 6 | 10
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6 | 16
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 14
Hypertension (Vascular disorders) | 5 | 8
Lymphocyte count decreased (Investigations) | 5 | 18
Depression (Psychiatric disorders) | 4 | 8
Influenza like illness (General disorders) | 4 | 8
Dysuria (Renal and urinary disorders) | 3 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The multisite consortium can publish any time after the data is collected and analyzed by FibroGen. The investigator can only publish after the multisite consortium publishes (or tries to publish and fails). FibroGen has 60 days to review a publication and can extend the embargo up to an additional 120 days (or 180 total).

DOCUMENTS (2):
  • Study Protocol (2022-05-16): https://cdn.clinicaltrials.gov/large-docs/93/NCT03941093/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-24): https://cdn.clinicaltrials.gov/large-docs/93/NCT03941093/SAP_001.pdf